CLINICAL TRIAL: NCT00721916
Title: Randomized Phase II Study of S-1, Oral Leucovorin, and Oxaliplatin Combination Therapy (SOL) Versus 5-FU, l-LV and Oxaliplatin Combination Therapy (mFOLFOX6) in Patients With Untreated Metastatic Colorectal Cancer
Brief Title: Randomized Phase II Study of SOL for Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Taiho10020390
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): SOL(The combination therapy of S-1, Leucovorin, and Oxaliplatin)
  Interventions: Drug: SOL(The combination therapy of S-1, Leucovorin, and Oxaliplatin)
- 2 (Active Comparator): mFOLFOX6(The combination therapy of 5-FU, l-LV and Oxaliplatin)
  Interventions: Drug: mFOLFOX6(The combination therapy of 5-FU, l-LV and Oxaliplatin)

INTERVENTIONS:
Drug: SOL(The combination therapy of S-1, Leucovorin, and Oxaliplatin) — L-OHP 85 mg/m2 iv. for 2 hr on day 1 of each 2 weeks cycle S-1 40-60 mg bid day 1～day 7 LV 25 mg bid day 1～day 7
  Arms: 1
Drug: mFOLFOX6(The combination therapy of 5-FU, l-LV and Oxaliplatin) — L-OHP 85 mg/m2 iv. for 2 hr on day 1 of each 2 weeks cycle l-LV 200 mg/m2 iv. for 2 hr on day 1 5-FU 400 mg/m2 bolus on day 1 5-FU 2400 mg/m2 ci for 46 hr (day 1, 2hr～48hr)
  Arms: 2

SUMMARY:
This is a randomized, multicenter study designed to evaluate the progression free survival of the SOL group (S-1, Leucovorin, and Oxaliplatin) compared with the mFOLFOX6 group (5-FU, l-LV and Oxaliplatin) as first-line treatment of patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved adenocarcinoma (colorectal cancer).
* Age: 20 ≤ at enrollment.
* No prior treatment (ex. radiation therapy, chemotherapy, hormonal therapy) to advanced disease. Patients who received adjuvant chemotherapy more than 180 days before enrollment can be allowed but those who received S-1 or Oxaliplatin containing treatment shall be excluded.
* At least one measurable lesion by RECIST criteria

Exclusion Criteria:

* Serious drug hypersensitivity.
* Prior history of peripheral neuropathy.
* Diarrhea .
* Simultaneously active double cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Until progression

SECONDARY OUTCOMES:
Safety | During chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Narikazu Boku, MD, Study Chair — St. Marianna University School of Medicine
Locations (1):
- Shizuoka Cancer Center, Shimonagakubo Nagaizumi-cho Sunto-gun, Shizuoka, Japan